CLINICAL TRIAL: NCT00571363
Title: A Randomised Study Comparing Tissue Conservation in Conventional Versus Mohs' Surgery of Basal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Responsible Party: Frank Muller, Specialist Registrar in Dermatology, NHS Tayside,
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2003DS10; R&D Project ID: 2003DS10
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Mohs Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard surgery (Active Comparator): basal cell carcinomas were excised with 4 mm margins
  Interventions: Procedure: standard surgery
- Mohs (Active Comparator): Basal cell carcinoma were removed via Mohs Micrographic surgery
  Interventions: Procedure: Mohs micrographic surgery

INTERVENTIONS:
Procedure: standard surgery — excision with 4 mm margins
  Arms: standard surgery
Procedure: Mohs micrographic surgery — excision of basal cell carcinoma with 2 mm margins and immediate examination of margins for residual tumour. residual tumour was excised until complete tumour removal was achieved.
  Arms: Mohs

SUMMARY:
We have compared to types of surgery to assess which one leaves the smaller surgical defect.

DETAILED DESCRIPTION:
Patients with a clinical diagnosis of a nodular basal cell carcinoma of less than 1 centimetre and 1 centimetre away from eyes, nose and ears were either randomized to undergo Mohs Micrographic Surgery or standard surgical excision. After the tumour had been removed the defect was measured.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of a nodular basal cell carcinoma of less than 1 cm, 1 cm away from eye, nose or ears

Exclusion Criteria:

* Subjects of less than 18 years of age
* Subjects unable to comply with instructions,
* Immunosuppressed subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
defect size after surgery | immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Muller, Principal Investigator — NHS Tayside
Locations (1):
- Ninewells Hospital and Medical School, Dundee, United Kingdom

REFERENCES:
- [Derived] Muller FM, Dawe RS, Moseley H, Fleming CJ. Randomized comparison of Mohs micrographic surgery and surgical excision for small nodular basal cell carcinoma: tissue-sparing outcome. Dermatol Surg. 2009 Sep;35(9):1349-54. doi: 10.1111/j.1524-4725.2009.01240.x. Epub 2009 Jun 3. PMID 19500127